CLINICAL TRIAL: NCT03596138
Title: Reliability and Reproducibility of Automated Angular Measurement in Strabismus
Acronym: FREGMA
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC18_0062
Record Dates: First submitted 2018-07-10; First posted 2018-07-23 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Strabismus
Keywords: angle measurement; automated; strabismus
MeSH Terms: conditions — Strabismus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Evaluate the reliability and reproductibility of the automated angular measurement by the Gazelab — Compare the results of the Gazelab to the alternate occlusion by prism bar (standard gold) examiners.

SUMMARY:
Angular measurement of deviation is an essential element in the clinical evaluation of strabic patients. It is performed by orthoptic methods. However, studies show that the same patient presents a great variability of his angular measurement between 2 consultations, and between 2 observers.

Automated angle measurement is a recent concept that aims to overcome the defects of subjective angle measurement by alternate occlusion test and prismatic bar.

Improvements made by these devices would provide reliable, objective and reproducible measurements of the angle of deviation by increasing the accuracy of strabal angle assessment, improving decision making and surgical follow-up, decreasing inter-examiner variability and variability over time, and facilitating data comparison to improve scientific publication possibilities.

The Gazelab® device is a video-oculograph combined with a laser projection system and an infrared camera. It allows an objective angular evaluation, in non-dissociating physiological conditions, possible even in the absence of binocular vision and allows an analysis of the deviation in all positions.

There is extremely little data in the literature on automated measuring devices. The Gazelab tool is still little known in the strabology discipline and seems to have a number of advantages over other devices. The interest of this examination towards this pathology led the ophthalmology department to use it in the current practice, and since recently it is an act nomenclaturé.

DETAILED DESCRIPTION:
The objective of this work is to evaluate the reliability and reproducibility of the automated angular measurement by the Gazelab® (ES12/13127) apparatus, compared to the standard gold which is the angular measurement by alternate occlusion test and prismatic bar, in horizontal strabisms (converging and diverging). Indeed in our daily practice the 2 examinations are carried out. To compare with the standard gold which denotes a strong inter-observer variability, the investigator will compare the results of the Gazelab to the alternate occlusion by prism bar (standard gold) 2 times with 2 trained examiners

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Strabic convergent or divergent patients or patients requiring an oculomotor check-up in their follow-up consultation
* Patient giving oral consent to this study

Exclusion Criteria:

* Patient with medical follow-up impossible,
* Impossibility to install Gazelab equipment for anatomical reasons of the head (craniostenosis...)
* No ocular fixation.
* Major without freedom under guardianship or trusteeship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Strabismus is a pathology that affects 2 to 4% of the French population. The Ophthalmology Department sees 200 adult patients with strabismus per month. In 6 months it will be easy to include in 30 months 30 patients of convergent strabismus and 30 of divergent strabismus. For patients with eye strain who do not have eye refractive errors the Department of Ophthalmology sees 2000 patients per month, to include these 30 patients in 6 months.
  Since this study is a prospective non-interventional research study, the patient may be part of a biomedical research study.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2019-04-29 (Actual); Study Completion 2019-04-29 (Actual)

PRIMARY OUTCOMES:
Intra-class correlation coefficient | 12 months
  Intra-class correlation coefficient calculated on the 4 measures (2 of each technique) of each patient taken at time 1 by the same assessor.

SECONDARY OUTCOMES:
Intra-class correlation coefficient using measurements | 12 months
  Intra-class correlation coefficient using measurements from each technique between 2 different evaluators at time 1
Intraclass correlation coefficient using time 1 and time 2 measurements | 12 months
  Intraclass correlation coefficient using time 1 and time 2 measurements with the same investigator

CONTACTS AND LOCATIONS:
Overall Officials: Pierre LEBRANCHU, Dr, Principal Investigator — Nantes University Hospital
Locations (1):
- CHU Nantes, Nantes, France